CLINICAL TRIAL: NCT00831974
Title: Phase IIa, Open-label, Randomized Study of Oral AB1010 in Patients With Systemic Indolent Mastocytosis With Handicap and Not Bearing Activating Point Mutations in the Phosphotransferase Domain of c-Kit Such as the Main Mutation Asp-816-Val (D816V)
Brief Title: Efficacy of AB1010 in Patients With Systemic Indolent Mastocytosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB04010
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Mastocytosis
Keywords: mastocytosis; indolent; handicap; wild-type; systemic; not D816V mutated
MeSH Terms: conditions — Mastocytosis | interventions — masitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): masitinib (AB1010) 6 mg/kg/day
  Interventions: Drug: masitinib (AB1010)
- 1 (Experimental): masitinib (AB1010) 3 mg/kg/day
  Interventions: Drug: masitinib (AB1010)

INTERVENTIONS:
Drug: masitinib (AB1010) — 3 mg/kg/day
  Arms: 1
Drug: masitinib (AB1010) — 6 mg/kg/day
  Arms: 2

SUMMARY:
This is a 12 weeks study aimed at assessing the safety and efficacy of 2 doses of AB1010 in patients suffering from indolent systemic mastocytosis with handicap.

DETAILED DESCRIPTION:
Efficacy will be assessed based on:

Pruritus score Number of flush per day Pollakyuria (on a daily basis) Number of stools per day QLQ-C30 score Hamilton Rating Scale for depression

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented Indolent systemic mastocytosis with handicap (ISMwh) having at least 2 infiltrated* organs (skin and /or bone-marrow and/or internal organ).
2. Bone-marrow, or skin or internal biopsy-documented mastocytosis and evaluable disease.
3. The absence of an activating point mutation in the phosphotransferase domain of c-Kit such as D816V c-Kit mutation in at least one of the two infiltrated organs: bone marrow and/or skin and/or other tissue.
4. Handicap defined as at least one of the following handicaps:

   * a number of flush per day ≥ 1 ,
   * a pruritus score ≥ 9 ,
   * a number of stools per day ≥ 4 ,
   * a Pollakyuria (on a per day basis) ≥ 8 ,
   * a QLQ-C30 score ≥ 83 ,
   * a Hamilton rating scale for depression ≥ 12

Exclusion Criteria:

1. Performance status > 2 (ECOG).
2. Inadequate organ function, except if the abnormalities are due to involvement by mast cells

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-10; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Response on: Pruritus score, Number of flush per day, Pollakyuria (on a daily basis), Number of stools per day, QLQ-C30 score, Hamilton Rating Scale for depression | 12 weeks

SECONDARY OUTCOMES:
AFIRMM score, reduction of organ infiltration,level of tryptase, reduction on bio markers (TNFα, eosinophils, histamine levels), pharmacokinetic profile of AB1010 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lortholary, MD, PhD, Principal Investigator — Hôpital Necker, Paris, France

REFERENCES:
- [Result] Paul C, Sans B, Suarez F, Casassus P, Barete S, Lanternier F, Grandpeix-Guyodo C, Dubreuil P, Palmerini F, Mansfield CD, Gineste P, Moussy A, Hermine O, Lortholary O. Masitinib for the treatment of systemic and cutaneous mastocytosis with handicap: a phase 2a study. Am J Hematol. 2010 Dec;85(12):921-5. doi: 10.1002/ajh.21894. PMID 21108325